CLINICAL TRIAL: NCT01149863
Title: WCI1680-09: Evaluation of Alterations in Time of Administration of Plerixafor (Mozobil ®, AMD3100) in Combination With G-CSF on Safety and CD34+ Cell Mobilization
Brief Title: Alteration in Timing of Plerixafor Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, R. Donald Harvey, PharmD, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00034057; WCI1680-09 (Other: Other)
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-05

CONDITIONS: Autologous Transplantation
Keywords: Autologous Transplantation
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plerixafor 17 hours prior to apheresis (Experimental): Dosing of plerixafor will occur at 3PM (1500 hours).
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor 240 mcg/kg SC will be administered daily starting on the first day of stem cell apheresis, up to a total of 4 doses.
  Other Names: AMD3100; Mozobil

SUMMARY:
Typically, the collection of blood cells for autologous stem cell transplant is done after the drugs granulocyte colony-stimulating factor (G-CSF) and plerixafor have been given to activate the bone marrow stem cells to produce a certain type of blood cell, called CD34+ cells. Currently, plerixafor is given in the evening, about 11 hours before apheresis (removal of blood) begins the following morning. The purpose of this study is to test whether plerixafor can instead be given 17 hours before apheresis. This timing would be more convenient since plerixafor would be given during normal clinic hours, and so patients would be within a clinic environment if any side effects develop.

The study will look for the activation of CD34+ cells in patients who receive plerixafor 17 hours before apheresis. We will follow the number of patients that achieve the target numbers of CD34+ cells, and the total number of CD34+ cells collected. These will be compared to the numbers in previous studies giving plerixafor 11 hours before apheresis.

We will also assess the safety of giving plerixafor 17 hours before apheresis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. MM patients in first or second complete or partial remission
3. ECOG performance status of 0 or 1
4. Up to 3 prior treatment regimens
5. Meet all eligibility requirements for autologous transplant
6. Adequate marrow function defined as WBC >3,000; ANC >1,500/mm3 ; Platelets >75,000/mm3
7. Adequate renal function defined as creatinine clearance > 30 mL/min by Cockcroft-Gault
8. Adequate liver function defined as AST/ALT/Bilirubin < 2 times upper limit of normal
9. Able to provide informed consent
10. Women not pregnant and agree to use contraception

Exclusion Criteria:

1. High risk co-morbidities for acute treatment complications (e.g., symptomatic coronary artery disease)
2. Brain metastases or carcinomatous meningitis
3. Previous treatment with high dose chemotherapy and autologous transplant.
4. Previous attempt to collect B-HPCs following mobilization with growth factors alone, growth factors and chemotherapy, or plerixafor and growth factors.
5. Acute infection or unexplained fever >38°C
6. Weight > 175% of ideal body weight as defined by the Devine equation.
7. Experimental therapy within 4 weeks
8. Cytokine administration in the previous 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Donald Harvey, PharmD, FCCP, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Plerixafor 17 Hours Prior to Apheresis: Dosing of plerixafor will occur at 3PM (1500 hours).
  Plerixafor : Plerixafor 240 mcg/kg SC will be administered daily starting on the first day of stem cell apheresis, up to a total of 4 doses.
Period: Overall Study
Arm/Group | Plerixafor 17 Hours Prior to Apheresis
Started | 34
Completed | 31
Not Completed | 3
Not completed — Missing data or Not receiveing studydrug | 3

BASELINE CHARACTERISTICS:
Arm/Group | Plerixafor 17 Hours Prior to Apheresis
Number analyzed (Participants) | 34
Age, Customized [Median (Full Range); unit: Years] | 59 [40 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Collected ≥ 6 x 10^6 CD34+ Cells by Day 5 (4 Apheresis Sessions) With Plerixafor Administration at 1500.
Time Frame: Within the first 5 days following plerixafor initiation
Measure: Number; unit: Participants
Arm/Group | Plerixafor 17 Hours Prior to Apheresis
Number analyzed (Participants) | 31
Participants | 31

2. Secondary Outcome: Number of Patients Who on Day 1 Collected > 10 x 10^6 CD34+ Cells/kg Following Plerixafor Dosing at 1500 Hrs
Time Frame: Within the first 5 days following plerixafor initiation
Measure: Number; unit: Participants
Arm/Group | Plerixafor 17 Hours Prior to Apheresis
Number analyzed (Participants) | 31
Participants | 22

ADVERSE EVENTS:
Arm/Group | Plerixafor 17 Hours Prior to Apheresis
Serious Adverse Events (participants affected / at risk) | 2/31
Other Adverse Events (participants affected / at risk) | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plerixafor 17 Hours Prior to Apheresis (N=31)
Hypokalemia (Blood and lymphatic system disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plerixafor 17 Hours Prior to Apheresis (N=31)
Bone Pain (Musculoskeletal and connective tissue disorders) | 16
Nausea (General disorders) | 11
Injection site reactions (Surgical and medical procedures) | 10
hypokalemia (Blood and lymphatic system disorders) | 7
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes